CLINICAL TRIAL: NCT05537636
Title: Effect of Regional Interdepence Physical Therapy Approach on Non-structural Medial Elbow Pain
Brief Title: Physical Therapy on Non-structural Medial Elbow Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Uhl (Other)
Collaborators: Bluegrass Orthopedics (Unknown)
Responsible Party: Sponsor-Investigator, Timothy Uhl, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60696
Record Dates: First submitted 2022-08-11; First posted 2022-09-13 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Elbow Injuries and Disorders; Neuritis, Ulnar; Neuritis, Brachial; Neuritis; Nerve Root; Neuritis Median Nerve
Keywords: Regional Interdependence; Posture; Neural Tension; Physical Therapy
MeSH Terms: conditions — Elbow Injuries; Disease; Ulnar Neuropathies; Brachial Plexus Neuritis; Neuritis | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Cohort longitudinal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regional Interdepence Intervention for the upper quarter (Experimental): Physical therapist will perform interventions to the entire uppper extremity and spine to treat elbow pain. Physical therapy intervention will include manual therapy and soft-tissue massage to the shoulder, cervical, and thoracic spine. Participants will be prescribed specific exercises using a phased approach.
  Interventions: Other: Rehabiltiation using exercise and manual therapy

INTERVENTIONS:
Other: Rehabiltiation using exercise and manual therapy — A licensed Physical Therapist will provide manual therapy to help restore spinal and scapular mobility. In association with this patients will be prescribed home exercises using a phased approach.
  Phase 1 to gain mobility of the spine and scapular motor control Phase 2 to gain shoulder mobility to strengthen scapular and spine musculature Phase 3 shoulder strengthening with long lever arms.

SUMMARY:
This study is investigating the effect of using a regional interdependence approach of managing non-structural elbow pain with physical therapy.

DETAILED DESCRIPTION:
Potential patients will be referred for physical therapy with elbow nerve pain arising from a non-structural lesion. We believe by addressing spine and trunk posture and mobility we can relieve elbow pain associated with a nerve compression with physical therapy.

Patients will be put on a staged exercise program to regain spinal mobility and strengthen proximal core musculature and scapular musculature. Manual therapy to facilitate mobility will be incorporated. Patients will undergo standard physical therapy by an unblinded therapist until resolution of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The patient presents with elbow pain that is not exacerbated with resisted wrist flexion, extension, supination, or pronation.
* The patient presents with elbow pain that is not exacerbated with passive wrist flexion or extension.
* The patient presents with three of the four positive cervical radicular signs
* Patient presents with peripheral paresthesia

Exclusion Criteria:

* The patient reports a surgical history involving the elbow.
* The patient has an MRI that is positive for structural deficits within the upper extremity.
* The patient self-reports a diagnosis of rheumatoid arthritis or other neurological systemic diseases such as Parkinson's disease, cerebrovascular accident, multiple sclerosis, or similar conditions

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Cervical Range of Motion in extension | Baseline and every 5th visit up to discharge which is estimated to be 3 months on average
  Inclinometer measurement of cervical extension
Change in Focus On Therapeutic Outcome (FOTO) Patient Outcme Score | Baseline and every 5th visit up to discharge which is estimated to be 3 months on average
  Patient self-report of perceived level of function. Scores range from 0 = low function, to 100=high function.
Change in Lower Trapezius scapular muscle strength | Baseline and every 5th visit up to discharge which is estimated to be 3 months on average
  Objectively measure with hand held dynamometer for scapular retraction

SECONDARY OUTCOMES:
Change in Elbow Flexion Range of Motion in Ulnar Nerve Tension position | Baseline and every 5th visit up to discharge which is estimated to be 3 months on average
  Goniometric measure using a standard plastic goniometer with patient plased In nerve tension position that bias tension on ulnar nerve. The standard upper limb tension test position described by Magee' Orthopaedic Physical Assessment 7th edition. The angle of elbow flexion that reproduces symptoms will be recorded. Values will range from 0-150 degrees with a higher numbers indicating less symptoms.
Change in Elbow Extension Range of Motion in Median Nerve Tension positoin | Baseline and every 5th visit up to discharge which is estimated to be 3 months on average
  Goniometric measure using a standard plastic goniometer with patient plased In nerve tension position that bias tension on median nerve. The standard upper limb tension test position described by Magee' Orthopaedic Physical Assessment 7th edition. The angle of elbow extension that reproduces symptoms will be recorded. Values will range from 0-150 degrees with a lower numbers indicating less symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tim L Uhl, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Bluegrass Orthopaedics, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sueki DG, Cleland JA, Wainner RS. A regional interdependence model of musculoskeletal dysfunction: research, mechanisms, and clinical implications. J Man Manip Ther. 2013 May;21(2):90-102. doi: 10.1179/2042618612Y.0000000027. PMID 24421619
- [Result] Wickstrom BM, Oakley PA, Harrison DE. Non-surgical relief of cervical radiculopathy through reduction of forward head posture and restoration of cervical lordosis: a case report. J Phys Ther Sci. 2017 Aug;29(8):1472-1474. doi: 10.1589/jpts.29.1472. Epub 2017 Aug 10. PMID 28878485
- [Result] Day JM, Willoughby J, Pitts DG, McCallum M, Foister R, Uhl TL. Outcomes following the conservative management of patients with non-radicular peripheral neuropathic pain. J Hand Ther. 2014 Jul-Sep;27(3):192-9; quiz 200. doi: 10.1016/j.jht.2014.02.003. Epub 2014 Feb 27. PMID 24685569
- [Result] Wainner RS, Fritz JM, Irrgang JJ, Boninger ML, Delitto A, Allison S. Reliability and diagnostic accuracy of the clinical examination and patient self-report measures for cervical radiculopathy. Spine (Phila Pa 1976). 2003 Jan 1;28(1):52-62. doi: 10.1097/00007632-200301010-00014. PMID 12544957
- [Result] Nee RJ, Jull GA, Vicenzino B, Coppieters MW. The validity of upper-limb neurodynamic tests for detecting peripheral neuropathic pain. J Orthop Sports Phys Ther. 2012 May;42(5):413-24. doi: 10.2519/jospt.2012.3988. Epub 2012 Mar 8. PMID 22402638